CLINICAL TRIAL: NCT06692309
Title: To Explore the Predictive Value of Electroencephalography Features in Perioperative Neurocognitive Disorders in Patients Undergoing Cardiovascular Surgery Under General Anaesthesia: a Single-centre Prospective Observational Study
Brief Title: Exploring the Predictive Value of Electroencephalography Features in Perioperative Neurocognitive Disorders Following Cardiovascular Surgery
Status: Recruiting | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DXK2022-ke-487
Record Dates: First submitted 2024-05-22; First posted 2024-11-18 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Surgery; Perioperative Neurocognitive Disorders
Keywords: Perioperative Neurocognitive Disorders;Electroencephalography
MeSH Terms: interventions — Cardiovascular Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Perioperative Neurocognitive Disorders: Postoperative delirium was assessed using the confusion assessment method or the confusion assessment method for the intensive care unit (CAM/CAM-ICU) .
  Cognitive levels were assessed 1 day before surgery and 1 week after surgery (7±2 days) using the Montreal Cognitive Assessment (MoCA). Patients were followed up one month (30±2 days) after surgery using the Telephone version of the Montreal Cognitive Assessment Scale (T-MoCA).
  Interventions: Procedure: cardiovascular surgery
- No-Perioperative Neurocognitive Disorders: Postoperative delirium was assessed using the confusion assessment method or the confusion assessment method for the intensive care unit (CAM/CAM-ICU) .
  Cognitive levels were assessed 1 day before surgery and 1 week after surgery (7±2 days) using the Montreal Cognitive Assessment (MoCA). Patients were followed up one month (30±2 days) after surgery using the Telephone version of the Montreal Cognitive Assessment Scale (T-MoCA).
  Interventions: Procedure: cardiovascular surgery

INTERVENTIONS:
Procedure: cardiovascular surgery — Heart bypass surgery; Heart valve replacement surgery

SUMMARY:
To explore the predictive value of Electroencephalography features in Perioperative Neurocognitive Disorders in patients undergoing cardiovascular surgery under general anesthesia

DETAILED DESCRIPTION:
Data was acquired on the ward using a 10-20 system with a standard 32-channel EEG cap and an EEG instrument (BP Company, Gilching, Germany). Patients were tested using cognitive assessment scales before and after surgery.

Cognitive levels were assessed 1 day before surgery and 1 week after surgery (7±2 days) using the Montreal Cognitive Assessment (MoCA) . Patients were followed up one month (30±2 days) after surgery using the Telephone version of the Montreal Cognitive Assessment Scale (T-MoCA).

Preoperative and postoperative electroencephalography brain network-related indexes (such as cluster coefficient, small world index, etc.) in patients with PND will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. undergoing coronary artery bypass surgery or valve replacement surgery under general anaesthesia
3. ASA grade: II-IV
4. older than 60 years
5. Able to complete cognitive function tests

Exclusion criteria:

1. history of severe neurological diseases and psychiatric diseases
2. history of drug abuse
3. severe hearing or vision impairment
4. preoperative delirium
5. serious adverse reactions such as cardiac arrest and cardiopulmonary resuscitation during surgery
6. patients undergoing secondary surgery in a short period
7. participation in concurrent clinical trials

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. older than 60 years
  2. ASA grade: I-III
  3. undergoing coronary artery bypass surgery or valve replacement surgery under general anaesthesia
  4. able to complete cognitive function tests
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
The predictive value of preoperative Electroencephalography features in patients with postoperative cognitive dysfunction following cardiovascular surgery | 2025.08
  Data was acquired on the ward using a 10-20 system with a standard 32-channel EEG cap and an EEG instrument (BP Company, Gilching, Germany). Patients were tested using cognitive assessment scales before and after surgery.
  Cognitive levels were assessed 1 day before surgery and 1 week after surgery (7±2 days) using The Montreal Cognitive Assessment (MoCA) . Patients were followed up one month (30±2 days) after surgery using the Telephone version of the Montreal Cognitive Assessment Scale (T-MoCA).

SECONDARY OUTCOMES:
The predictive value of preoperative Electroencephalography features in patients with postoperative delirium following cardiovascular surgery | 2025.08
  Postoperative delirium was assessed using the confusion assessment method or the confusion assessment method for the intensive care unit (CAM/CAM-ICU) .
Electroencephalography features in patients with postoperative delirium | 2025.08
  Electroencephalography was collected in delirium patients one week(7±2 days) after surgery. Postoperative delirium was assessed using the confusion assessment method or the confusion assessment method for the intensive care unit (CAM/CAM-ICU) .
  Preoperative and postoperative electroencephalography brain network-related indexes (such as cluster coefficient, small world index, etc.) in patients with postoperative delirium will be included in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anshi Wu, doctor, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided